CLINICAL TRIAL: NCT03709186
Title: Radiomic Markers for Breast Cancer Metastasis Using Dynamic Contrast Enhanced MRI and Diffusion-Weighted MRI
Brief Title: Radiomic Markers for Breast Cancer Metastasis and Treatment Response Using MRI
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. William Tran, Radiation Therapist Clinician Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: 214-2018
Record Dates: First submitted 2018-10-12; First posted 2018-10-17 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2019-10

CONDITIONS: Invasive Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary aim of the study is to identify radiomic features as biomarkers of metastatic progression following primary therapy.

DETAILED DESCRIPTION:
The study aims to evaluate radiomic markers in breast tumors to evaluate metastatic risk based on radiomic features following primary therapy. The investigators aim to analyze images at various time intervals before, during and after primary treatments using two advanced imaging techniques (DCE-MRI & DWI-MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must give appropriate written informed consent prior to participation in the study;
2. Subjects must be able and willing to comply with the safety procedures during the scanning period;
3. Subjects must be men and women age 18+
4. Biopsy-confirmed diagnosis of invasive breast cancer; (ER+/-, PR+/-, HER2+/-).
5. Stage I-III disease according to the AJCC v7 criteria.
6. Patients with sufficient renal function (creatinine clearance, i.e., >=30 mL/min/1.73 m2).
7. Primary treatments can include neoadjuvant chemotherapy or surgery

Exclusion Criteria:

* 1. Subjects with a past medical history of abnormalities, significant injury, or medical or surgical procedures (e.g. Silicone/saline implants) involving either breast, exclusive of the lesion at issue.

  2. Subjects with any dermatologic abnormalities (including tattoos, open sores, or breached skin) involving either breast 3. Subjects with a current or past medical history of connective tissue disease 4. Subjects who are pregnant or lactating 5. Subjects with an implanted electronic device such as a cardiac pacemaker, defibrillator, or neurological stimulator 6. Subjects, who, in the opinion of the investigator or clinical research coordinator, may not otherwise be appropriate for inclusion into the study, such as significant anxiety, history of musculoskeletal disease which may predispose them to discomfort during the imaging/scanning period.

  7. Allergies to any contrast agent administered to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enrol women and men with a pathologically-confirmed diagnosis of invasive breast cancer that is stage I-III according to the AJCC v7 criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) | Up to 60 months
  Evaluating the degree of absence of residual cancer cells

SECONDARY OUTCOMES:
Time to distant breast cancer recurrence (months) | Up to 60 months
  Evaluating the time until a recurrence event has occurred in the breast.
Time to distant metastasis | Up to 60 months
  Evaluating onset of distant metastasis
Time to death | Up to 60 months
  Evaluating time to cancer-related death

CONTACTS AND LOCATIONS:
Overall Officials: William T. Tran, MRT(T), PhD, Principal Investigator — Radiation Therapist Clinician Scientist; Colleen Bailey, PhD, Principal Investigator — Sunnybrook Research Institute; Angus Lau, PhD, Principal Investigator — Sunnybrook Research Institute; Kasia Jerzak, MD, MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada